CLINICAL TRIAL: NCT00882882
Title: A Relative Bioavailability Study of Metformin HCL 500 mg XR Tablets Under Fasting Conditions
Brief Title: To Demonstrate the Relative Bioavailability of Metformin HCL 500 mg Extended Release (XR) Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B013701
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-04

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

ARMS (4):
- 1 (Experimental): Metformin HCL 500 mg Extended-Release Tablets, Geneva PTC
  Interventions: Drug: Metformin HCL 500 mg Extended-Release Tablets, Geneva PTC
- 2 (Experimental): Metformin HCL 500 mg Extended-Release Tablets, Geneva PTC
  Interventions: Drug: Metformin HCL 500 mg Extended-Release Tablets, Geneva PTC
- 3 (Active Comparator): GLUCOPHAGE XR 500 mg Extended-Release Tablets Bristol-Myers Squibb
  Interventions: Drug: GLUCOPHAGE XR 500 mg ER Tablets Bristol-Myers Squibb
- 4 (Active Comparator): GLUCOPHAGE XR 500 mg Extended-Release Tablets Bristol-Myers Squibb
  Interventions: Drug: GLUCOPHAGE XR 500 mg ER Tablets Bristol-Myers Squibb

INTERVENTIONS:
Drug: Metformin HCL 500 mg Extended-Release Tablets, Geneva PTC
  Arms: 1
Drug: Metformin HCL 500 mg Extended-Release Tablets, Geneva PTC
  Arms: 2
Drug: GLUCOPHAGE XR 500 mg ER Tablets Bristol-Myers Squibb
  Arms: 3
Drug: GLUCOPHAGE XR 500 mg ER Tablets Bristol-Myers Squibb
  Arms: 4

SUMMARY:
To demonstrate the relative bioavailability of Metformin HCl 500 mg XR tablets under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2001-06; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 23 days

CONTACTS AND LOCATIONS:
Overall Officials: So Ran Hong, M.D., Principal Investigator — Novum Independent Institutional Review Board